CLINICAL TRIAL: NCT01620580
Title: Symptom Management Program for Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Francess Danquah, Assistant Professor, Nursing, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-SN-11-0465
Record Dates: First submitted 2011-10-24; First posted 2012-06-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Haemodialysis-induced Symptom
Keywords: sleep disturbance; tiredness; itching & numbness
MeSH Terms: conditions — Parasomnias; Fatigue; Pruritus; Hypesthesia | interventions — Self-Management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self Management Strategies (Active Comparator): Participants in the intervention group will receive printed self management strategies each of the 5 symptoms, a symptom diary with the self-management strategies and a 15 minutes discussion. The intervention script will instruct participants on how to use the printed strategies by PI and RA #1.
  Week 3.
  Interventions: Behavioral: Self-management
- Dietary Information (Active Comparator): Control arm
  Interventions: Behavioral: Dietary Information

INTERVENTIONS:
Behavioral: Self-management — Participants in the intervention group will receive printed self management strategies each of the 5 symptoms, a symptom diary with the self-management strategies and a 15 minutes discussion. The intervention script will instruct participants on how to use the printed strategies by PI and RA #1.
  Week 3
  Other Names: Behavioral
  Arms: Self Management Strategies
Behavioral: Dietary Information — The control or usual care group will receive a symptom diary designed for the control group without any strategies and a 5 minutes discussion on how to complete the diary from RA# 1. The PI will make weekly follow up calls on the same schedule as the intervention group starting week 4 until week 7 for a total of 4 calls focusing on enhancing healthy eating skills & adherence to renal diet and fluid restriction without discussing any intervention with the group.
  Other Names: Behavioral
  Arms: Dietary Information

SUMMARY:
Self-management intervention may decrease symptom burden and improve functioning over time.

DETAILED DESCRIPTION:
Self-management intervention (strategies) may decrease symptom burden (sleep disturbance, tiredness; itching and numbness) and improve functioning (social, physical and emotional) over time(baseline, 3 weeks and 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years old,
2. on HD three times a week,
3. received HD for ≥ six months,
4. read and write English,
5. have telephone service.

Exclusion Criteria:

* history of dementia,
* acquired immunodeficiency syndrome (AIDS) and active cancer, and
* inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Decrease symptom burden | 8 weeks
  The study aims are:
  1. To compare the differences between the self management intervention and control group on the following outcomes:
  1. Decreased symptoms: itching, tiredness, numbness, sleep disturbance (difficulty falling asleep & difficulty staying asleep);
  2. Adherence to treatment diary Improved social functioning, physical functioning and emotional status.

SECONDARY OUTCOMES:
Feasibility of implementing self management intervention | 5 weeks
  To evaluate the feasibility of implementing the self management intervention for a larger randomized controlled studyTreatment delivered (number of interventions sessions delivered and strategies used); Treatment receipts (understanding of strategies); and Treatment enactment (reported perception of usefulness of the strategies).

CONTACTS AND LOCATIONS:
Overall Officials: Francess V Danquah, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - DaVita Summit Dialysis, Houston, Texas
  - DaVita Houston Dialysis, Houston, Texas

REFERENCES:
- [Background] Dodd M, Janson S, Facione N, Faucett J, Froelicher ES, Humphreys J, Lee K, Miaskowski C, Puntillo K, Rankin S, Taylor D. Advancing the science of symptom management. J Adv Nurs. 2001 Mar;33(5):668-76. doi: 10.1046/j.1365-2648.2001.01697.x. PMID 11298204
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264